CLINICAL TRIAL: NCT06153329
Title: An Open-label, Active-controlled, Randomized, Three-cycle, Crossover Trial to Evaluate the Pharmacokinetics and Pharmacodynamics of Single-Dose THDB0206 Injection in Healthy Chinese Subjects
Brief Title: A Trial to Evaluate the Pharmacokinetics and Pharmacodynamics of THDB0206 Injection in Healthy Chinese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tonghua Dongbao Pharmaceutical Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: THDB0206L04
Record Dates: First submitted 2023-11-17; First posted 2023-12-01 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Healthy
MeSH Terms: interventions — Insulin Lispro

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- THDB0206 injection (Experimental)
  Interventions: Drug: THDB0206 injection
- Humalog® (Active Comparator)
  Interventions: Drug: Humalog®
- BC222insulin lispro injection (Active Comparator)
  Interventions: Drug: BC222insulin lispro injection

INTERVENTIONS:
Drug: THDB0206 injection — 0.2 U/kg, single-dose administration, subcutaneous injection 5 cm laterally from the belly button on the left or right side of the abdominal wall
  Arms: THDB0206 injection
Drug: Humalog® — 0.2 U/kg, single-dose administration, subcutaneous injection 5 cm laterally from the belly button on the left or right side of the abdominal wall
  Arms: Humalog®
Drug: BC222insulin lispro injection — 0.2 U/kg, single-dose administration, subcutaneous injection 5 cm laterally from the belly button on the left or right side of the abdominal wall
  Arms: BC222insulin lispro injection

SUMMARY:
This is a single-center, single-dose, open-label, positive-controlled, randomized, three-cycle, crossover 8-hour euglycemic clamp study to evaluate the PK, PD, safety and tolerability of THDB0206 injection after subcutaneous injection in healthy Chinese subjects. This trial will enroll 39 subjects to receive the investigational medicinal products.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who provide a signed and dated informed consent form (Appendix 1) before starting any study-related activities (study-related activities are any procedures that will not be involved during the normal management of subjects).
2. Healthy local Chinese males or females, who complete medical history, physical examination and laboratory tests according to the judgment of the investigator.
3. Aged ≥ 18 years and ≤ 40 years when signing the informed consent form.
4. Body mass index (BMI) ≥ 18 kg/m2 and < 25 kg/m2 at screening, male weight ≥ 50 kg, female weight ≥ 45 kg.
5. Intravenous fasting blood glucose < 6.1 mmol/L and intravenous blood glucose < 7.8 mmol/L 2 hours after the glucose load in the 75 g oral glucose tolerance test at screening.
6. According to local laboratory analysis, glycated hemoglobin HbA1c≤6.1% st screening.

Exclusion Criteria:

Subjects who meet any of the following criteria will be excluded from the study:

1. Known or suspected allergies to investigational medicinal products and related products, or a history of multiple and/or severe allergies to drugs or food.
2. Subjects who have previously participated in this study (participation in the study is defined as randomization), or received any drugs in the clinical development stage within 3 months before the screening of this study.
3. Any cancer or history of cancer, including basal cell skin cancer or squamous cell skin cancer.
4. According to the judgment of the investigator, any clinically relevant cardiovascular, respiratory, gastrointestinal, liver, kidney, metabolism, endocrine, hematology (bleeding diseases), skin, venereal disease, nervous system, mental disease or other major diseases or related medical history.
5. During the screening visit, abnormal values of hematology, blood biochemistry, blood coagulation or urinalysis have clinical significance, and the investigator judges and considers potential diseases.
6. According to the judgment of the investigator, the results of the insulin release test has clinically significant abnormalities at screening.
7. Heart problems, defined as the presence of decompensated heart failure (New York Heart Association Class III and IV) at any time and/or angina pectoris within 12 months prior to screening and/or acute myocardial infarction at any time.
8. According to the judgment of the investigator, the blood pressure has clinically significant abnormalities at screening.
9. The heart rate detected by 12-lead ECG at rest exceeds the range of 50-100 beats per minute (including 50 and 100 beats).
10. According to the judgment of the investigator, the standard 12-lead ECG has clinically significant abnormalities at screening.
11. Increased risk of thromboembolism, such as known coagulopathy, (family) history of thrombosis, related arrhythmias (e.g., paroxysmal atrial fibrillation), etc.
12. Mental disorders or language barriers which prevent full understanding or cooperation.
13. According to the investigator's judgment, there is a history of deep vein thrombosis in the lower extremities or a first-degree relative (parents, siblings or children) frequently develops deep vein thrombosis in the lower extremities.
14. Any disease or condition that the investigator believes will pose an unacceptable risk to the safety of the subjects.
15. Subjects who have used any drugs (prescription drugs and over-the-counter drugs) within 14 days before administration of the IMP or within 5 times the elimination half-life of the IMP (whichever is longer).
16. According to the investigator's judgment, subjects with a history of alcoholism or drug/chemical drug abuse, or subjects with positive drug screening/breath alcohol test results during the screening visit, or subjects drinking more than 21 units of alcohol per week (male subjects) or 14 units of alcohol (female subjects) (1 unit of alcohol is equivalent to approximately 330 mL of beer, 1 glass of 120 mL of wine or 40 mL of spirits).
17. Subjects who have smoked more than 5 cigarettes per day on average within one year before the screening visit and do not agree to quit smoking during the study period.
18. Female subjects who have a positive pregnancy test result during the screening visit or on Day -1 of Visit 2.
19. According to the diagnostic test used locally, hepatitis B surface antigen or hepatitis C antibody is positive (or active hepatitis is diagnosed according to local practice), or human immunodeficiency virus (HIV) antibody test result is positive, or syphilis test result is positive.
20. Subjects who have donated blood or plasma in the past month, or donated more than 300 mL within 3 months before the screening visit.
21. During the period from the first administration to the end of the study, male subjects who are sexually active and have not been sterilized, and their female partners who are still fertile, the subjects themselves and their partners not using effective contraceptive measures (effective contraceptive measures mean methods that have an unintended pregnancy rate of less than 1% each year, including surgical sterilization, condoms, intrauterine device (birth control ring), abstinence).
22. Women of childbearing age who are pregnant, breastfeeding, preparing for pregnancy, and have not used effective contraceptive measures, or postmenopausal women who have had less than 1 year of amenorrhea and serum follicle stimulating hormone (FSH) level ≤ 40 IU/L and have not used effective contraceptive measures.
23. During the COVID-19 pandemic period, those who have lived or traveled in areas with a high incidence of COVID-19, have contact history with confirmed or suspected infected people, have a history of fever clinic visits, or those who are positive for the COVID-19 nucleic acid test/positive for the new coronavirus seroantibodies.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2021-06-17 (Actual); Primary Completion 2022-06-06 (Actual); Study Completion 2022-06-06 (Actual)

PRIMARY OUTCOMES:
AUCLisp(0-30 min) | From 0 to 30 minutes
  Area under the insulin lispro plasma concentration-time curve from 0 to 30 minutes

SECONDARY OUTCOMES:
Cmax (Lisp) | From 0 to 8 hours
  The maximum plasma concentration of insulin lispro observed
AUCLisp | From 0 to 8 hours
  Area under the insulin lispro plasma concentration-time curve
tmax(Lisp) | From 0 to 8 hours
  Time to reach the maximum insulin lispro plasma concentration
t1/2 | From 0 to 8 hours
  Terminal half-life
CL/F | From 0 to 8 hours
  Apparent clearance
Vz/F | From 0 to 8 hours
  Apparent volume of distribution
AUCGIR | From 0 to 8 hours
  Area under the glucose infusion rate-time curve
GIRtot | From 0 to 8 hours
  Total glucose infusion during clamping
GIRmax | From 0 to 8 hours
  Maximum glucose infusion rate
tGIRmax | From 0 to 8 hours
  Time to reach the maximum glucose infusion rate
Number of participants with abnormal clinical laboratory findings (haematology, biochemistry and urinalysis) | From the first drug administration to the follow-up visit (3 to 10 days after the last drug administration)
Number of participants with abnormal 12-lead ECG parameters (PR, QR, QRS intervals and QTc) | From the first drug administration to the follow-up visit (3 to 10 days after the last drug administration)
Number of participants with abnormal vital signs (body temperature, supine blood pressure and pulse rate) | From the first drug administration to the follow-up visit (3 to 10 days after the last drug administration)
Number of participants with abnormal physical examination (general condition, head and five sense organs, neck, chest, abdomen, spine and limbs, nervous system) | From the first drug administration to the follow-up visit (3 to 10 days after the last drug administration)
Number of participants with hypoglycemia events in each treatment arm | From the first drug administration to the follow-up visit (3 to 10 days after the last drug administration)
Number of participants with injection site reactions (spontaneous pain, tenderness, itching, redness, edema, induration/infiltration) | From the first drug administration to the follow-up visit (3 to 10 days after the last drug administration)
Number of participants with AE and SAE | From the first drug administration to the follow-up visit (3 to 10 days after the last drug administration)

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital of Sichuan University, Sichuan, China

IPD SHARING:
Plan to Share IPD: No